CLINICAL TRIAL: NCT03797651
Title: Ticagrelor Monotherapy in PAtients Treated With New-generation Drug-eluting Stents for Acute Coronary Syndrome; T-PASS Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0782
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease, Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard DAPT (Active Comparator): Patient will continue standard treatment (aspirin plus ticagrelor) for 1 year. Dosage of ticagrelor would be 90 mg twice a day, and 100 mg of aspirin will be prescribed once a day.
  Interventions: Drug: Standard DAPT
- Very-short DAPT within 1 month (Experimental): Patient will stop aspirin after discharge (DAPT less than 1 months after PCI) (ticagrelor monotherapy). Dosage of ticagrelor would be 90 mg twice a day, and 100 mg of aspirin will be prescribed once a day (during hospitalization).
  Interventions: Drug: Very-short DAPT less than 1 month after PCI

INTERVENTIONS:
Drug: Standard DAPT — Patient will continue standard treatment (aspirin plus ticagrelor) for 1 year. Dosage of ticagrelor would be 90 mg twice a day, and 100 mg of aspirin will be prescribed once a day.
  Arms: Standard DAPT
Drug: Very-short DAPT less than 1 month after PCI — Patient will stop aspirin (ticagrelor monotherapy) after discharge or within 1 month. Dosage of ticagrelor would be 90 mg twice a day, and 100 mg of aspirin will be prescribed once a day (during hospitalization).
  Arms: Very-short DAPT within 1 month

SUMMARY:
We hypothesized that ticagrelor monotherapy might be enough to prevent thromboembolic events without aspirin after PCI in patients with acute coronary syndrome(ACS). Moreover, ticagrelor monotherapy will reduce bleeding risk compared to DAPT with aspirin plus ticagrelor. We will also evaluate 1-year safety and efficacy of Orsiro stent for patient with acute coronary syndrome. After confirmation of enrollment, patients will be randomized to continue standard treatment (aspirin plus ticagrelor) for 1 year or to stop aspirin after discharge or less than 1 month after PCI (ticagrelor monotherapy). Randomization will be stratified according to 1) the presence of diabetes and 2) ST elevation myocardial infarction (MI). Baseline clinical and angiographic characteristics, laboratory findings will be assessed at the time of randomization. All patients will provide informed consent on their own initiative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥19 years old
2. Patients who received new generation sirolimus-eluting (Orsiro® series) stent implantation for treating ACS, including acute MI and unstable angina
3. Provision of informed consent

Exclusion Criteria:

1. Age> 80 years
2. Increased risk of bleeding, anemia, thrombocytopenia
3. A need for oral anticoagulation therapy
4. Pregnant women or women with potential childbearing
5. Life expectancy < 1 year

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2850 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Net clinical benefit | 1 year after procedure
  A composite of all-cause death, MI, stent thrombosis, stroke, major bleeding

SECONDARY OUTCOMES:
Each components of net clinical benefit | 1 year after procedure
  All-cause death, MI, stent thrombosis, stroke, major bleeding
Cardiovascular mortality | 1 year after procedure
  Cardiovascular mortality
Major or minor bleeding | 1 year after procedure
  Major or minor bleeding
Major adverse cardiac event | 1 year after procedure
  A composite of cardiac death, MI, stent thrombosis, ischemia-driven target-vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Myeong-Ki Hong, Principal Investigator — Division of Cardiology, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei Cardiovascular Center and Cardiovascular Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong SJ, Lee SJ, Suh Y, Yun KH, Kang TS, Shin S, Kwon SW, Lee JW, Cho DK, Park JK, Bae JW, Kang WC, Kim S, Lee YJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; T-PASS (Ticagrelor Monotherapy in Patients Treated With New-Generation Drug-Eluting Stents for Acute Coronary Syndrome) Investigators. Stopping Aspirin Within 1 Month After Stenting for Ticagrelor Monotherapy in Acute Coronary Syndrome: The T-PASS Randomized Noninferiority Trial. Circulation. 2024 Feb 20;149(8):562-573. doi: 10.1161/CIRCULATIONAHA.123.066943. Epub 2023 Oct 25. PMID 37878786